CLINICAL TRIAL: NCT05910034
Title: The Study of Envafolimab Plus Docetaxel in Combination With or Without Trilaciclib Versus Docetaxel in Advanced NSCLC Previously Treated With a PD-1 Inhibitor Combined With Chemotherapy
Brief Title: Envafolimab Plus Docetaxel In Combination With or Without Trilaciclib Versus Docetaxel in Advanced NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, professor of medicine, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMA-NSCLC-012
Record Dates: First submitted 2023-06-10; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: Trilaciclib; Envafolimab; NSCLC; Second-line Treatment
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trilaciclib+Envafolimab+Docetaxel (Experimental): Trilaciclib:240mg/m2 IV d1,within 4h before chemotherapy; Envafolimab:300mg SC d1,Q3W; Docetaxel:75mg/m2 IV d1, Q3W
  Interventions: Drug: Trilaciclib+Envafolimab+Docetaxel
- Envafolimab+Docetaxel (Experimental): Envafolimab:300mg SC d1,Q3W; Docetaxel:75mg/m2 IV d1, Q3W
  Interventions: Drug: Envafolimab+Docetaxel
- Docetaxel (Experimental): Docetaxel: 75mg/m2 IV d1, Q3W
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Trilaciclib+Envafolimab+Docetaxel — This is a multi-arm, randomized, controlled, multicenter, Phase II clinical study. Participants randomly assigned at a 1:1:1 ratio to three groups, and will be treated until disease progression, intolerance, withdrawal of consent or completion determined by the investigator.
  Arms: Trilaciclib+Envafolimab+Docetaxel
Drug: Envafolimab+Docetaxel — This is a multi-arm, randomized, controlled, multicenter, Phase II clinical study. Participants randomly assigned at a 1:1:1 ratio to three groups, and will be treated until disease progression, intolerance, withdrawal of consent or completion determined by the investigator.
  Arms: Envafolimab+Docetaxel
Drug: Docetaxel — This is a multi-arm, randomized, controlled, multicenter, Phase II clinical study. Participants randomly assigned at a 1:1:1 ratio to three groups, and will be treated until disease progression, intolerance, withdrawal of consent or completion determined by the investigator.
  Arms: Docetaxel

SUMMARY:
To evaluate the efficacy and safety of Envafolimab Plus Docetaxel in combination with or without Trilaciclib versus docetaxel IN patients with advanced non-small cell lung cancer previously treated with a PD-1 inhibitor combined with chemotherapy

DETAILED DESCRIPTION:
Trilaciclib indication: Trilaciclib, a CDK4/6 inhibitor, was used before chemotherapy to reduce the incidence of bone marrow suppression, approved by FDA and NMPA for small cell lung cancer in 2021 and in 2022.

Envafolimab indication: Envafolimab, a PD-L1 inhibitor, was used for unresectable or metastatic, MSI-H or dMMR, Adult patients with advanced solid tumors, approved by NMPA in 2021.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged≥ 18 years old
* Metastatic or advanced (stage IV) NSCLC confirmed by tissue or pathology
* Patients with advanced NSCLC who had previously failed treatment with platinum-containing chemotherapy combined with PD-1 inhibitor
* Disease must be measurable by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).,and has at least one measurable lesion
* Patients with asymptomatic brain metastasis or whose symptoms are stable after treatment
* Patients who responded to initial therapy or whose disease was stable for at least 3 months
* Laboratory tests met the following criteria:

  1. Hemoglobin (Hb)≥100 g/L(female), ≥110g/L(male)
  2. Neutrophils (ANC)≥1.5×109/L
  3. platelet count (PLT)≥100×109/L
  4. Cr≤ 15mg/L or CrCl≥ 60 mL/min
  5. TBIL≤ 1.5×ULN
  6. ALT and AST ≤ 3 × ULN or ≤5× ULN(patients with liver metastases)
  7. Albumin ≥ 30 g/L
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1
* Estimated life expectancy of more than 12 weeks
* Women: All women with potential fertility must have negative serum pregnancy tests during the screening period and must have reliable contraception after signing the informed consent form until 3 months after the last dose
* Already signed an informed consent form

Exclusion Criteria:

* Diagnosis of other malignancies than NSCLC within 5 years prior to the first dose administration (excluding radically treated cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and/or radically resected carcinoma in situ)
* Toxicity not recovered to ≤ Grade 1 from prior anticancer therapy
* Previous treatment with PD-L1 inhibitors
* ≥grade 3 immune-related adverse reactions have occurred during previous PD-1 inhibitors treatment
* Patients with known or suspected interstitial pneumonia
* Patients with known positive driving genes(EGFR,ALK,ROS1)
* Have used or requirement of treatment with prednisone > 10 mg/day or equivalent systemic corticosteroids within 14 days prior to the first dose of study drug
* Administration of live attenuated vaccines within 28 days prior to the first study drug treatment or planned administration during the study
* Uncontrolled ischemic heart disease or clinically significant congestive heart failure (NYHA grade III or IV)
* Have stroke or cardiovascular events within 6 months prior to enrollment
* QTcF>480 msec or QTcF>500 msec(patients with ventricular pacemakers)
* Patients who have received hematopoietic stem cell or bone marrow transplants
* Allergic to the study drug or its ingredients
* Any other circumstances in which the researcher believes that the patient is not suitable to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 12 months after the last subject participating in
  Progression-free survival (PFS per RECIST 1.1) is defined as the time from randomization to the date of first documentation of disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
ORR | 12 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) in total subjects.
DCR | 12 months after the last subject participating in
  The proportion of subjects with complete response (CR), partial response (PR)and stable disease in(SD) in total subjects.
DoR | 12 months after the last subject participating in
  DoR (per RECIST 1.1) is defined as the time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.
OS | 24 months after the last subject participating in
  Defined as the time from randomization to all-cause death.
QOL | 24 months after the last subject participating in
  Quality of life was assessed using the EQ-5D-5L scale
The incidence of Subjects With Treatment-Emergent Adverse Events (TEAEs) According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 | 24 months after the last subject participating in
  TEAEs will be defined as the adverse events (AEs) that occur between first dose of study drug administration and 28 days after the last dose of study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jialei, doctor, Study Chair — Fudan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morimoto Y, Kishida T, Kotani SI, Takayama K, Mazda O. Interferon-beta signal may up-regulate PD-L1 expression through IRF9-dependent and independent pathways in lung cancer cells. Biochem Biophys Res Commun. 2018 Dec 9;507(1-4):330-336. doi: 10.1016/j.bbrc.2018.11.035. Epub 2018 Nov 14. PMID 30446226
- [Result] Travis WD, Brambilla E, Nicholson AG, Yatabe Y, Austin JHM, Beasley MB, Chirieac LR, Dacic S, Duhig E, Flieder DB, Geisinger K, Hirsch FR, Ishikawa Y, Kerr KM, Noguchi M, Pelosi G, Powell CA, Tsao MS, Wistuba I; WHO Panel. The 2015 World Health Organization Classification of Lung Tumors: Impact of Genetic, Clinical and Radiologic Advances Since the 2004 Classification. J Thorac Oncol. 2015 Sep;10(9):1243-1260. doi: 10.1097/JTO.0000000000000630. PMID 26291008
- [Result] Boyero L, Sanchez-Gastaldo A, Alonso M, Noguera-Ucles JF, Molina-Pinelo S, Bernabe-Caro R. Primary and Acquired Resistance to Immunotherapy in Lung Cancer: Unveiling the Mechanisms Underlying of Immune Checkpoint Blockade Therapy. Cancers (Basel). 2020 Dec 11;12(12):3729. doi: 10.3390/cancers12123729. PMID 33322522
- [Result] Herbst RS, Garon EB, Kim DW, Cho BC, Gervais R, Perez-Gracia JL, Han JY, Majem M, Forster MD, Monnet I, Novello S, Gubens MA, Boyer M, Su WC, Samkari A, Jensen EH, Kobie J, Piperdi B, Baas P. Five Year Survival Update From KEYNOTE-010: Pembrolizumab Versus Docetaxel for Previously Treated, Programmed Death-Ligand 1-Positive Advanced NSCLC. J Thorac Oncol. 2021 Oct;16(10):1718-1732. doi: 10.1016/j.jtho.2021.05.001. Epub 2021 May 26. PMID 34048946
- [Result] Law AMK, Valdes-Mora F, Gallego-Ortega D. Myeloid-Derived Suppressor Cells as a Therapeutic Target for Cancer. Cells. 2020 Feb 27;9(3):561. doi: 10.3390/cells9030561. PMID 32121014
- [Result] Cabrita R, Mitra S, Sanna A, Ekedahl H, Lovgren K, Olsson H, Ingvar C, Isaksson K, Lauss M, Carneiro A, Jonsson G. The Role of PTEN Loss in Immune Escape, Melanoma Prognosis and Therapy Response. Cancers (Basel). 2020 Mar 21;12(3):742. doi: 10.3390/cancers12030742. PMID 32245160
- [Result] Roselli M, Cereda V, di Bari MG, Formica V, Spila A, Jochems C, Farsaci B, Donahue R, Gulley JL, Schlom J, Guadagni F. Effects of conventional therapeutic interventions on the number and function of regulatory T cells. Oncoimmunology. 2013 Oct 1;2(10):e27025. doi: 10.4161/onci.27025. PMID 24353914